CLINICAL TRIAL: NCT01022437
Title: Geranium Oil and Its Components for the Relief of Numbness-OB 100
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Clinical Medical Doctor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PBRC 28041
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Nerve Conduction; Numbness
MeSH Terms: conditions — Hypesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Geranium Oil and component PN-34 (Experimental)
  Interventions: Other: Geranium Oil with component PN-34

INTERVENTIONS:
Other: Geranium Oil with component PN-34 — Geranium oil as a topical application to the body that is numb, time to determine how long it takes for the feeling to return, if it does so, and if the return of feeling is maintained by daily topical application of oil over 12 weeks. This including the process of absorption, distribution and localization.

SUMMARY:
This study is designed to evaluate the effectiveness of geranium oil and its components in the relief of numbness and the restoration of sensations.

DETAILED DESCRIPTION:
This is a pilot study to define the time course, the incidence of sensation restoration and the improvement in nerve conduction in people with numbness by using topical geranium oil.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Neuropathy with the inability to feel touch in a standard nylon filament test
* Signed informed consent

Exclusion Criteria:

* Pregnant or nursing
* Known allergies to geranium oil or geranium oil fractions
* Open sore in the area of numbness
* Migraine headaches or headaches to strong smells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response to numbness relief and restoration of sensation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alok Gupta, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Penningto Biomedical Research Center, Baton Rouge, Louisiana, United States